CLINICAL TRIAL: NCT04013594
Title: Effect of Preoperative Oral Carbohydrates on the Glycemic Variability of Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2019-0428
Record Dates: First submitted 2019-06-26; First posted 2019-07-09 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- carbohydrate group(CHO group) (Experimental)
  Interventions: Dietary Supplement: carbohydrate group
- control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: carbohydrate group — Randomly selected patients of the carbohydrate group are given oral carbohydrate (400ml) 2-3 hours before surgery.
  Arms: carbohydrate group(CHO group)

SUMMARY:
Preoperative carbohydrate drink intake attenuate insulin resistance. However, carbohydrate loading may compromise blood glucose control in patients with diabetes. There is some evidence that oral carbohydrate loading may be safe in patients with type 2 diabetes. Therefore, the investigators aim to evaluate whether preoperative carbohydrate intake affects insulin resistance and glycemic variability in patients with diabetes. Fifty patients scheduled for total knee arthroplasty will be divided into carbohydrate (n=25) and control (n=25) groups. Randomly selected patients of the carbohydrate group are given 400ml of 12.8 g/100 ml carbohydrate beverage 2-3 hours before their scheduled operation. In contrast, patients in the control group are fasted from water 2 hours before surgery according to standard protocol.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing total knee arthroplasty

Exclusion Criteria:

* 1. Patients with contraindications to spinal anesthesia (local infection, clotting disorders, anatomical abnormalities, sepsis, etc.)
* 2. Patients with gastroesophageal reflux disease, gastric emptying disorders, inflammatory bowel disease, or previous treatment for intra-abdominal cancer
* 3. Patients with chronic renal disease or severe cardiovascular disease
* 4. HbA1c >69 mmol/mol or BMI >30 kg/m2
* 5. A duration of ≥5 hours between consumption of CHO and initiation of surgery.
* 6. The subject is a foreigner or illiterate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2020-10-07 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Glycemic variability | Before anesthesia
  - Coefficient of glucose variability =SD/mean x 100 (%)
Glycemic variability | Before anesthesia
  - J index=0.001 x (MBG +SD)2 mg/dL
Glycemic variability | immediately after anesthesia
  - Coefficient of glucose variability =SD/mean x 100 (%)
Glycemic variability | immediately after anesthesia
  - J index=0.001 x (MBG +SD)2 mg/dL
Glycemic variability | operation end
  - Coefficient of glucose variability =SD/mean x 100 (%)
Glycemic variability | operation end
  - J index=0.001 x (MBG +SD)2 mg/dL
Glycemic variability | 1 hour after surgery
  - Coefficient of glucose variability =SD/mean x 100 (%)
Glycemic variability | 1 hour after surgery
  - J index=0.001 x (MBG +SD)2 mg/dL

SECONDARY OUTCOMES:
Insulin resistance | Before anesthesia
  Insulin resistance index = fasting glucose x fasting insulin/22.5
Insulin resistance | Before anesthesia
  serum laboratory test: glucagon
Insulin resistance | Before anesthesia
  serum laboratory test: GLP-1
Insulin resistance | Before anesthesia
  serum laboratory test: C-peptide
Insulin resistance | Before anesthesia
  serum laboratory test: free fatty acid
gastric volume | Before anesthesia
  gastric volume measured by ultrasonography.
hand grip strength | Before anesthesia
  hand grip strength measured by electronic hand dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Soop M, Nygren J, Myrenfors P, Thorell A, Ljungqvist O. Preoperative oral carbohydrate treatment attenuates immediate postoperative insulin resistance. Am J Physiol Endocrinol Metab. 2001 Apr;280(4):E576-83. doi: 10.1152/ajpendo.2001.280.4.E576. PMID 11254464
- [Background] Gustafsson UO, Nygren J, Thorell A, Soop M, Hellstrom PM, Ljungqvist O, Hagstrom-Toft E. Pre-operative carbohydrate loading may be used in type 2 diabetes patients. Acta Anaesthesiol Scand. 2008 Aug;52(7):946-51. doi: 10.1111/j.1399-6576.2008.01599.x. Epub 2008 Mar 7. PMID 18331374
- [Derived] Lee B, Kim SY, Cho BW, Suh S, Park KK, Choi YS. Preoperative Carbohydrate Drink Intake Increases Glycemic Variability in Patients with Type 2 Diabetes Mellitus in Total Joint Arthroplasty: A Prospective Randomized Trial. World J Surg. 2022 Apr;46(4):791-799. doi: 10.1007/s00268-021-06437-1. Epub 2022 Jan 10. PMID 35006328